CLINICAL TRIAL: NCT07404371
Title: Efficacy of Sensory Reweighting Techniques for Balance and Risk of Fall in Chronic Ischemic Stroke Patients
Acronym: SRT-IS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montiha Azeem (Other)
Responsible Party: Sponsor-Investigator, Montiha Azeem, Principal investigator, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/15/03/30
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Ischemic Stroke
Keywords: Sensory Reweighting; Balance Training; Fall Risk

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A Sensory Reweighting Balance Training Group (Experimental): Participants in this arm will receive sensory reweighting-based balance training aimed at enhancing integration of visual, vestibular, and somatosensory inputs for postural control. The intervention will be delivered three times per week for eight weeks, with each session lasting approximately 45 minutes. Training will include balance tasks performed under altered sensory conditions such as reduced visual input, compliant surfaces, head movements, and dual-task activities. Exercise difficulty will be progressively increased according to individual tolerance while ensuring participant safety.
  Interventions: Behavioral: Sensory Reweighting Balance Training
- group B Conventional Balance Training Group (Active Comparator): Participants in this arm will receive conventional balance training without sensory reweighting components. The program will be delivered three times per week for eight weeks, with each session lasting approximately 45 minutes. Exercises will focus on static and dynamic balance tasks, including standing with a narrow base, sit-to-stand practice, and forward/backward walking. No manipulation of sensory input will be included. Training intensity and duration will be matched to the experimental group to allow fair comparison of outcomes.
  Interventions: Behavioral: Conventional Balance Training

INTERVENTIONS:
Behavioral: Sensory Reweighting Balance Training — Participants will receive sensory reweighting-based balance training aimed at improving postural control by enhancing the central nervous system's ability to integrate visual, vestibular, and somatosensory inputs. Training will be conducted three times per week for eight weeks, with 45-minute sessions including warm-up, core balance exercises, and cool-down. Exercises will be performed under altered sensory conditions, such as standing on foam surfaces, performing tasks with eyes closed, head movements during stance and gait, and dual-task activities. Task difficulty will be progressively increased based on individual tolerance while maintaining safety.
  Arms: group A Sensory Reweighting Balance Training Group
Behavioral: Conventional Balance Training — Participants will receive conventional balance training without sensory reweighting components. The program will be delivered three times per week for eight weeks, with each session lasting approximately 45 minutes. Exercises will focus on static and dynamic balance tasks such as standing with a narrow base, sit-to-stand practice, and forward/backward walking. No manipulation of sensory input will be included. Training intensity and duration will be matched to the experimental group to ensure comparability of outcomes.
  Arms: group B Conventional Balance Training Group

SUMMARY:
This randomized controlled trial will evaluate the effectiveness of sensory reweighting techniques on balance and risk of falls in individuals with chronic ischemic stroke. A total of 46 participants will be recruited using purposive sampling and randomly assigned into two groups through the sealed envelope method. Balance and fall risk will be assessed using the Berg Balance Scale and the Timed Up and Go test at baseline and after completion of the intervention. Participants in the experimental group will receive sensory reweighting-based balance training three times per week for eight weeks, incorporating altered sensory conditions such as reduced visual input, unstable surfaces, and vestibular challenges. The control group will receive conventional balance training of similar duration and intensity without sensory manipulation. Both groups will also receive standard physiotherapy throughout the intervention period. Ethical approval will be obtained prior to data collection, written informed consent will be secured from all participants, and confidentiality and voluntary participation will be ensured.

DETAILED DESCRIPTION:
This study will be conducted as a randomized controlled trial to investigate the efficacy of sensory reweighting techniques in improving balance and reducing the risk of falls among patients with chronic ischemic stroke. Following ethical approval, participants will be recruited from selected rehabilitation centers using a non-probability purposive sampling technique. A total of 46 eligible participants, including an allowance for dropout, will be enrolled and randomly allocated into experimental and control groups using the sealed envelope method to ensure unbiased group assignment. Individuals aged 40-60 years with a stroke duration of more than six months, adequate cognitive function, and the ability to stand and walk with or without assistive devices will be included.

Baseline data will be collected prior to intervention using standardized outcome measures. Balance performance will be assessed using the Berg Balance Scale, a validated tool consisting of 14 functional tasks that evaluate postural control and balance during daily activities. Risk of falls will be measured using the Timed Up and Go test, which assesses functional mobility by recording the time taken to stand from a chair, walk a short distance, turn, return, and sit down. Demographic and clinical information such as age, gender, duration of stroke, use of assistive devices, and fall history will also be documented.

Participants allocated to the experimental group will undergo a structured sensory reweighting balance training program aimed at enhancing the central nervous system's ability to integrate visual, vestibular, and somatosensory inputs for postural control. The intervention will be administered three times per week for eight weeks, with each session lasting approximately 45 minutes. Training will include balance tasks performed under progressively challenging sensory conditions, such as standing on compliant surfaces, performing tasks with eyes closed, incorporating head movements during stance and gait, and engaging in dual-task activities. Exercise intensity and task complexity will be gradually increased according to individual tolerance while maintaining participant safety.

Participants in the control group will receive conventional balance training with the same frequency and duration as the experimental group. This program will focus on traditional static and dynamic balance exercises, including standing with a narrowed base of support, sit-to-stand practice, and forward and backward walking. No manipulation of sensory input will be included in this group, allowing comparison between standard balance rehabilitation and sensory reweighting-based training.

In addition to group-specific interventions, all participants will receive standard physiotherapy throughout the study period. This will include passive and active range of motion exercises, functional strengthening, and gait training tailored to individual needs. Standard therapy will be delivered at moderate intensity for 20-25 minutes per session, five days per week, to ensure uniform baseline rehabilitation across both groups. Written informed consent will be obtained from all participants, confidentiality will be maintained, participation will be voluntary, and individuals will be free to withdraw from the study at any time without affecting their standard care.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed case of chronic ischemic stroke (duration >6 months post-stroke) Both male and female patients with age range 40-60 years . Able to stand and walk at least 10 feet (with or without assistive devices). Mini-Mental State Examination (MMSE) score ≥24 (to ensure adequate cognitive ability to follow instructions).

Medically stable and cleared by a physician to participate in balance training. Experiencing balance impairment and/or history of at least one fall in the past 6 months

Exclusion Criteria:

Hemorrhagic stroke patients or mixed stroke types Severe visual, auditory, or vestibular impairments not correctable by aids (which would interfere with sensory reweighting assessment).

Other neurological conditions (e.g., Parkinson's disease, multiple sclerosis, peripheral neuropathy).

Musculoskeletal disorders significantly affecting balance (e.g., recent fracture, severe arthritis).

On medications that severely affect balance or cause dizziness (e.g., sedatives, high-dose antiepileptic.

Severe aphasia or communication disorders impeding participation in the intervention

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-18 (Estimated)

PRIMARY OUTCOMES:
Balance Performance | Baseline and 8 weeks post-intervention
  Balance will be measured using the Berg Balance Scale (BBS), a validated clinical tool consisting of 14 functional tasks assessing postural control, stability, and fall risk in chronic ischemic stroke patients. Each task is scored from 0 (unable to perform) to 4 (independent and safe), with a maximum total score of 56. Higher scores indicate better balance, and scores below 45 suggest increased risk of falls. Assessments will be conducted at baseline and after completion of the 8-week intervention to evaluate the efficacy of sensory reweighting balance training compared to conventional balance exercises.

SECONDARY OUTCOMES:
Risk of Falls | Baseline and 8 weeks post-intervention
  Risk of falls will be evaluated using the Timed Up and Go (TUG) test, a standardized and widely used measure of functional mobility and dynamic balance in neurological populations. The test records the time (in seconds) required for a participant to stand up from a chair, walk 3 meters, turn around, walk back, and sit down. Shorter completion times indicate better mobility and lower fall risk, while times greater than 20 seconds suggest an increased risk of falls. The TUG test will be administered at baseline and after completion of the 8-week intervention to compare changes between the sensory reweighting training group and the conventional balance training group.

CONTACTS AND LOCATIONS:
Overall Officials: Kanwal Mirani, MSPTN, Principal Investigator — The University of Lahore, Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Lahore, Punjab Province, Pakistan